CLINICAL TRIAL: NCT03184740
Title: Physical Performance and Analgesic Effects of tDCS in Primary Dysmenorrhea: A Randomized, Double Blind Clinical Trial
Brief Title: Physical Performance and Analgesic Effects of tDCS in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Edson meneses da silva filho, Master student, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.530.846
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Transcranial Direct Current Stimulation; Dysmenorrhea Primary; Pain; Mental Disorders; Physical Fitness
MeSH Terms: conditions — Pain; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-tDCS (Experimental): A constant current (anodic) of 2mA will be applied for 20 minutes over the Primary motor cortex (M1).
  Interventions: Device: Active Transcranial Direct Current Stimulation
- Sham-tDCS (Sham Comparator): A constant current (sham) of 2mA will be applied on the Primary motor cortex, but the stimulator will be turned off after 30 seconds .
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — For electrode placement, the criteria used by the 10/20 electroencephalography system will be obeyed and the electrodes will be positioned over Primary motor cortex, C3 area for the anode and Fp2 (contralateral supraorbital area) for the cathode electrode. A constant current of 2mA will be applied for 20 minutes.
  Arms: Active-tDCS
Device: Sham Transcranial Direct Current Stimulation — For electrode placement, the criteria used by the 10/20 electroencephalography system will be obeyed and the electrodes will be positioned over primary motor cortex, C3 area for the anode and Fp2 (contralateral supraorbital area) for the cathode electrode, but the stimulator will be turned off after 30 seconds of stimulation.
  Arms: Sham-tDCS

SUMMARY:
Technological advances and non-invasive techniques to modulate brain function have been developed, including transcranial Direct Current Stimulation (tDCS). Basically, electrodes are placed on the brain regions to stimulate or inhibit it. Subsequently, a continuous electrical current (0.4-2 mA) is imposed, for a period of 3-20 minutes, to modify cortical excitability. Few are the research groups that work on the topic of primary dysmenorrhea and the use of tDCS as the focus of study. Preliminary studies associated the use of tDCS with pain reduction, but the outcomes of physical and behavioral function needs further investigation.

ELIGIBILITY:
Inclusion Criteria:

- to have primary dysmenorrhea symptoms for more than 6 months with a mean perception of at least 3 (on a scale of 0 to 10) on the visual analogue scale, to have a regular menstrual cycle from 28 to 32 days.

Exclusion Criteria:

- Participants will be excluded if they have history of genitourinary disease (infectious oncology or infection), neurogenic bladder dysfunction, to have alcohol or drug abuse in the last 6 months, to have severe depression (score greater than 30 on the Beck depression inventory), to have previously neurological disorders diagnosis and to be pregnant.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain | It will be used throughout the first and second menstrual cycle (approximately 60 days).
  Pain diary will be used to assess pain levels
Changes in pain | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Visual Analogue Scale will be used to measure pain levels
Changes in anxiety levels | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Hamilton anxiety rating scale will be used to measure anxiety levels
Changes in affectivity | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Positive And Negative Affect Scale will be used to measure affectivity
Changes in local pain levels | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Digital pressure algometry will be used to measure local pain levels
Changes in hand strength | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Hydraulic hand dynamometer will be used to measure hand strength
Changes in functional capacity | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Six-minute walk test will be used to measure functional capacity
Changes in flexibility | First evaluation will be done between the first and third days of initial menstrual cycle. The second evaluation will be done between the first and third days of the next menstrual cycle
  Thomas test will be used to measure flexibility

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Santa Cruz, Rio Grande do Norte, Brazil